CLINICAL TRIAL: NCT06912776
Title: Novel Visual Education Tool to Improve Recognition and Reporting of Postpartum Urgent Maternal Warning Signs
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Kaitlyn Neumann, Principal Investigator, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: STU00222375
Record Dates: First submitted 2025-03-27; First posted 2025-04-06 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Postpartum
Keywords: Pregnancy; Postpartum; nulliparus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Participant will view a visual aid picture (appendix A) first (Other): Participant will view a visual aid picture (appendix A) of a post delivery complication first.
  Interventions: Other: Participant will view a visual aid picture (appendix A) first
- Participant will view a visual aid picture (appendix B) first (Other): Participant will view a visual aid picture (appendix B) of a post delivery complication first
  Interventions: Other: Participant will view a visual aid picture (appendix B) first

INTERVENTIONS:
Other: Participant will view a visual aid picture (appendix A) first — Participant will view a visual aid picture (appendix A) of a post delivery complication first
  Arms: Participant will view a visual aid picture (appendix A) first
Other: Participant will view a visual aid picture (appendix B) first — Participant will view a visual aid picture (appendix B) of a post delivery complication first
  Arms: Participant will view a visual aid picture (appendix B) first

SUMMARY:
This study aims to create a novel visual education tool that builds on the urgent maternal warning signs identified by The Council on Patient Safety in Women's Health Care. Including effective images will improve the understanding of these grave warning signs/symptoms, improving anatomical accuracy while remaining simplistic for patients of varying levels of health care literacy. The investigative team will be focusing on urgent warning signs pertinent to the postpartum period.

ELIGIBILITY:
Inclusion Criteria:

* Postpartum women
* Nulliparity
* Age >18 years of age
* English speaking patients

Exclusion Criteria:

* Inability to provide informed written consent
* Refusal to participate in all study-related procedures
* Patients not fluent in English
* Patients with current or history of serious peripartum complications and/or events - such as DVT, PE, peripartum cardiomyopathy, etc. (in which the patient may have received more than standard clinical counseling)
* Patient with comorbidities that potentially require anticoagulation i.e. coagulopathies and may be more prone to DVTs
* Patients with uncorrected visual or hearing impairment
* Healthcare providers (in which patients will have significant background knowledge)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 40 (Estimated)
Dates: Start 2025-06-20 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Number of participants who recognize deep vein thrombosis, | 1 Day
  Participant will accurately identify the health care issue shown to participants and identified as Picture A and Picture B

SECONDARY OUTCOMES:
Number of participants who demonstrate understanding deep vein thrombosis, | 1 Day
  Participants written response of the understanding of deep vein thrombosis.
Number of participants who would report deep vein thrombosis | 1 Day
  After review of Picture A and Picture B number of participants who report deep vein thrombosis to their care provider or emergency room.

CONTACTS AND LOCATIONS:
Overall Officials: Kaitlyn Neumann, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern Medicine, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] You WB, Wolf MS, Bailey SC, Grobman WA. Improving patient understanding of preeclampsia: a randomized controlled trial. Am J Obstet Gynecol. 2012 May;206(5):431.e1-5. doi: 10.1016/j.ajog.2012.03.006. Epub 2012 Mar 13. PMID 22542120
- [Background] Delp C, Jones J. Communicating information to patients: the use of cartoon illustrations to improve comprehension of instructions. Acad Emerg Med. 1996 Mar;3(3):264-70. doi: 10.1111/j.1553-2712.1996.tb03431.x. PMID 8673784
- [Background] Houts PS, Bachrach R, Witmer JT, Tringali CA, Bucher JA, Localio RA. Using pictographs to enhance recall of spoken medical instructions. Patient Educ Couns. 1998 Oct;35(2):83-8. doi: 10.1016/s0738-3991(98)00065-2. PMID 10026551
- [Background] Burger G. SOAP Newsletter. 1998;Winter:6-9
- [Background] Council on Patient Safety in Women's Health Care. Urgent Maternal Warning Signs. May 2020, <https://safehealthcareforeverywoman.org>.